CLINICAL TRIAL: NCT03213795
Title: Anatomical Feasibility of Multibranched Off-the-shelf Endografts for Thoracoabdominal and Para-renal Aortic Aneurysms (TAMBE Study)
Acronym: TAMBE
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Principal Investigator, IRCCS San Raffaele
Other Study IDs: TAMBE/39/OSR
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Thoracoabdominal Aneurysms and Para-renal Aortic Aneurysms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Since the development of multibranched endografts a novel therapeutic option for the management of thoracoabdominal and para-renal aortic aneurysms was made accessible. The introduction of readily available off-the-shelf devices expanded the application of such technology also to those patients who could not afford to wait for a customized endograft to be designed and manufactured according to their aneurysm morphology

DETAILED DESCRIPTION:
To evaluate the theoretical anatomical feasibility of multibranched off-the-shelf endografts in patients with thoracoabdominal and para-renal aortic aneurysms based on retrospective review of pre-operative imaging studies of the patients treated for this pathology in the San Raffaele Hospital's Vascular Surgery Unit in the past ten years.

Materials and methods:

The investigators review retrospectively the pre-operative contrast-enhanced computed tomography scans (CTA), stored in the hospital PACS, of the 562 patients treated at the San Raffaele Hospital's Vascular Surgery Unit, between January 2007 and January 2017 by means of open aortic aneurysm repair. All patients involved in the study have already signed informed consent for data collection and analysis at hospital admission.

Inclusion criteria:

• patient who underwent treatment of thoracoabdominal or para-renal aortic aneurysm at San Raffaele Hospital in between January 2007 and January 2017.

Exclusion criteria:

• incomplete or inappropriate imaging quality defined as pre-operative CTAs with slice thickness >1-mm.

All preoperative CTAs with 1-mm slice thickness will be included in the study and analyzed on the dedicated workstation with OsiriX software (Pixmeo sarl, Bernex, Switzerland) currently employed in the Unit for imaging assessment.

Sensitive patient information will not be available during data analysis.

Vascular access will be evaluated according to the following inclusion criteria:

1. femoral and iliac artery diameter ≥8mm (24Fr) on one side and ≥5mm (16Fr) on the contralateral side, without severe calcification or tortuosity;
2. at least one patent vessel for anterograde branch cannulation (branchial/axillary/subclavian artery) with diameter ≥3mm.

The proportion of patients excluded due to inadequate vascular accesses will be reported in the final results together with diameter of the smallest access vessels determining the exclusion.

The selected patient sample will be subdivided in three groups:

1. extensive TAAA: including Crawford extent I and II TAAA;
2. Crawford extent III TAAA;
3. supra-renal aortic aneurysms: including Crawford extent IV TAAA and para-renal abdominal aortic aneurysms.

The latest 100 consecutive cases per group will be subsequently studied in order to assess the feasibility of an off-the-shelf endovascular approach.

Multi-planar and curved reconstruction of each patient CTA will be analyzed and the following measurements recorded using the top of the ostium of the celiac trunk as reference point:

1. patency of the target vessels (CT, SMA, LRA and RRA);
2. presence of accessory renal arteries or independent origin of celiac trunk branches;
3. inner diameter of the target vessels;
4. target vessels with aberrant or early branching, aneurysm or dissection, with <15mm of healthy artery for bridging stent placement;
5. radial orientation of the target vessels ("clock position", expressed in degrees);
6. orientation of the target vessels with respect to the longitudinal aortic axis (expressed in degrees);
7. distance to the top of the ostium of target vessels;
8. distance to aortic bifurcation and bilateral iliac bifurcation;
9. aneurysmatic involvement of common iliac arteries (max diameter >20mm);
10. distance to proximal aneurysm neck (25mm of healthy aorta);
11. distance to left subclavian artery;
12. inner and outer diameter at proximal neck, at 1cm and 2cm above proximal neck, at aortic bifurcation, and at common iliac artery bilaterally;
13. residual aortic lumen at CT, SMA and renal arteries emergence.

The feasibility will be evaluated considering the patients and endografts characteristics and all the technical steps required for a proper endovascular aneurysm exclusion.

All the assessed variables will be prospectively recorded in a Microsoft Office Excel database.

The clinical study will be carried out according to the ethical principles of the Declaration of Helsinki and following the active regulations on observational studies.

Analysis:

The extracted data will be employed to feed three major lines of research:

1. to evaluate the anatomical suitability of the novel investigational Gore TAMBE (W.L. Gore & Associates, Flagstaff, AZ, USA) multibranched off-the-shelf stent-graft for total endovascular management of thoracoabdominal and para-renal aortic aneurysms;
2. to evaluate the anatomical suitability, according to Instruction for Use and literature recommendations, of the commercially available Cook T-Branch (Cook Medical, Bloomington, IN, USA) multibranched off-the-shelf stent-graft for total endovascular management of thoracoabdominal and para-renal aortic aneurysms. This line of research will focus on the evaluation of the expected length of healthy aorta sacrificed to obtain appropriate proximal endograft sealing;
3. to compare the applicability of Gore TAMBE and Cook T-Branch endografts in TAAA of different extents and para-renal aneurysms.

The results of the three studies will be submitted for publication in peer-reviewed scientific journals focused on the field of vascular and endovascular surgery.

ELIGIBILITY:
Inclusion criteria:

• patient who underwent treatment of thoracoabdominal or para-renal aortic aneurysm at San Raffaele Hospital in between January 2007 and January 2017.

Exclusion criteria:

• incomplete or inappropriate imaging quality defined as pre-operative CTAs with slice thickness >1-mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient who underwent treatment of thoracoabdominal or para-renal aortic aneurysm at San Raffaele Hospital in between January 2007 and January 2017.
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
anatomical feasibility of multibranched off-the-shelf endografts in patients with thoracoabdominal and para-renal aortic aneurysms | 2007-2017
  evaluate the theoretical anatomical feasibility of multibranched off-the-shelf endografts in patients with thoracoabdominal and para-renal aortic aneurysms based on retrospective review of pre-operative imaging studies of the patients treated for this pathology in our Unit in the past ten years

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chuter TA, Rapp JH, Hiramoto JS, Schneider DB, Howell B, Reilly LM. Endovascular treatment of thoracoabdominal aortic aneurysms. J Vasc Surg. 2008 Jan;47(1):6-16. doi: 10.1016/j.jvs.2007.08.032. Epub 2007 Nov 5. PMID 17980540
- [Result] Sobocinski J, d'Utra G, O'Brien N, Midulla M, Maurel B, Guillou M, Azzaoui R, Roeder B, Resch TA, Haulon S. Off-the-shelf fenestrated endografts: a realistic option for more than 70% of patients with juxtarenal aneurysms. J Endovasc Ther. 2012 Apr;19(2):165-72. doi: 10.1583/11-3772.1. PMID 22545880
- [Derived] Cambiaghi T, Grandi A, Bilman V, Melissano G, Chiesa R, Bertoglio L. Anatomic feasibility of the investigational GORE EXCLUDER Thoracoabdominal Branch Endoprosthesis (TAMBE), off-the-shelf multibranched endograft for the treatment of pararenal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2021 Jan;73(1):22-30. doi: 10.1016/j.jvs.2020.03.056. Epub 2020 Apr 28. PMID 32360681